CLINICAL TRIAL: NCT06606288
Title: Characterizing Outcomes and Real-World Experience of Cardiac Physiologic Pacing (The CORE-CPP Study)
Acronym: CORE-CPP
Status: Active, not recruiting | Type: Observational
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Other Study IDs: 30489333
Record Dates: First submitted 2024-09-18; First posted 2024-09-23 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2024-09

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Conduction system pacing: Medicare beneficiaries indicated for CRT implanted with a Medtronic dual-chamber transvenous pacemaker on or after the study start date with lead type and placement data indicating conduction system pacing.
  Interventions: Device: Conduction system pacing
- Bi-ventricular pacing: Medicare beneficiaries indicated for CRT implanted with a Medtronic bi-ventricular pacemaker (CRT-P) on or after the study start date with lead type and placement data not indicating conduction system pacing.
  Interventions: Device: Bi-ventricular pacing

INTERVENTIONS:
Device: Conduction system pacing — Implant with a Medtronic dual-chamber transvenous pacemaker on or after the study data with lead type and placement data indicating conduction system pacing
  Groups: Conduction system pacing
Device: Bi-ventricular pacing — Implant with a Medtronic bi-ventricular pacemaker (CRT-P) on or after the study date
  Groups: Bi-ventricular pacing

SUMMARY:
The purpose of this study is to use real-world evidence to validate that conduction system pacing (CSP), delivered via a Medtronic 3830 catheter-delivered lead and a Medtronic dual-chamber transvenous pacemaker, is a safe and effective alternative to biventricular pacing (BVP) in patients indicated for cardiac resynchronization therapy (CRT) to deliver cardiac physiologic pacing (CPP), as documented in the clinical literature.

ELIGIBILITY:
Inclusion Criteria:

Dual-chamber CSP cohort:

* Medicare beneficiaries implanted with a Medtronic dual-chamber transvenous pacemaker on or after the study start date.
* Lead type and placement data indicating CSP.
* An indication for CRT.

BVP comparator cohort:

* Medicare beneficiaries implanted with a Medtronic biventricular pacemaker (CRT-P) on or after the study start date.

Exclusion Criteria:

Dual-chamber CSP cohort:

* Evidence of a prior CIED device.
* Less than 12 months continuous enrollment in Medicare Part A and Part B prior to implant date.
* Non-Medtronic pacemaker (unable to link to Medtronic device registration data).
* Missing lead type or placement data.
* Lead type and placement data indicating non-CSP placement.

BVP comparator cohort:

* Evidence of a prior CIED device.
* Less than 12 months continuous enrollment in Medicare Part A and Part B prior to implant date.
* Non-Medtronic pacemaker (unable to link to Medtronic device registration data).
* Missing lead type or placement data.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study cohort will include all U.S. Medicare beneficiaries enrolled in fee-for-service Medicare implanted with a Medtronic pacemaker between January 1, 2017 and December 1, 2023.
Sampling Method: Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Acute complication rate | 30 days
  Demonstrate that dual-chamber CSP is non-inferior to BVP on implant safety in patients indicated for CRT.
  Endpoint: Compare the acute (≤ 30 days) overall complication rate associated with dual chamber CSP vs. BVP. The acute overall complication rate is a composite measure of separate elements of complications (embolism and thrombosis, events at puncture site, cardiac effusion and perforation, device-related complications, and other procedural complications) and reinterventions (lead-related reinterventions, device revisions, replacements, removals, and upgrades to CRT).
Heart Failure Hospitalization Rate | 12 months
  Demonstrate that dual-chamber CSP is non-inferior to BVP in patients indicated for CRT.
  Endpoint: Compare the heart failure hospitalization rate associated with CSP vs. BVP in the CRT-indicated population.

SECONDARY OUTCOMES:
Device-Related Reintervention Rate | 12 months
  Compare the device-related reintervention rate associated with dual chamber CSP vs. BVP.
Heart Failure-All-Cause Mortality Composite | 12 months
  Compare the composite endpoint of heart failure hospitalization or all-cause mortality rate associated with dual=chamber CSP use vs. BVP in the CRT-indicated population.
All-Cause Mortality Rate | 12 months
  Compare the all-cause mortality rate associated with dual-chamber CSP use vs. BVP in the CRT-indicated population.

CONTACTS AND LOCATIONS:
Locations (1):
- Medtronic, Mounds View, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No
Sharing individual participant data is not permitted under the data use agreement with the Centers for Medicare and Medicaid Services (CMS) which allows us to access the Medicare data for research purposes.